CLINICAL TRIAL: NCT02486159
Title: The Oligonucleotide Chip Analysis for Allergic Rhinitis Treatment in Herbal Plaster and Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 98-0938B
Record Dates: First submitted 2015-06-16; First posted 2015-07-01 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2015-06

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Herbal plaster and Acupuncture (Experimental): In the first year: Acupoint herbal plaster applications every one week over a 4-week period for a total of 4 applications.
  In the second year: Acupoint herbal plaster used as the same method as first year, and combined with Acupuncture treatment in the same time.
  Interventions: Drug: Herbal plaster (Sanfujiu); Procedure: Acupuncture

INTERVENTIONS:
Drug: Herbal plaster (Sanfujiu) — The Acupoint herbal plaster consisted of mustard seed, fumarate, asarum, angelica, cinnamon, and ginger at a ratio of 3:3:2:2:0.5:4, respectively. The treatment was prepared by dissolving the ginger in water and adding the powder to form a plaster. Mixtures were formed into cakes of approximately 1.5 × 1.5 × 0.5 cm3 and were held in position using plastic sheets.
  Other Names: Sanfujiu
Procedure: Acupuncture — Eight (8) acupuncture treatment sessions over 4 weeks were performed for each volunteer. The standard protocol for acupuncture treatment covered the most commonly treated acupoints for allergic rhinitis: LI4, ST36, LI20 in both sides, and EX-HN3. After insertion of needles at each acupoint, manual stimulation of needles on LI20 and EX-HN3 was repeated 3 times at 5-minute intervals. Electrostimulation was applied to the needles inserted in ST36 and LI4 with a frequency of 3-5 Hz, and the intensity was adjusted according to each volunteer's tolerance. All needles were removed 20 minutes later in each treatment session.

SUMMARY:
Using Oligonucleotide Chip Analysis, investigators compared gene expression levels in allergic rhinitis patients before and after a series of acupoint herbal plaster and Acupuncture treatment.

In the first year, Twenty-three participants with persistent allergic rhinitis each received four acupoint herbal plaster treatments, applied using the moxibustion technique, and clinical outcomes were evaluated using the Rhinitis Quality of Life Questionnaire (RQLQ). Peripheral blood samples were analyzed using an ImmunoCAP Phadiatop test, and patients were classified as phadiatop (Ph)-positive or -negative. Microarray results were examined for genes that were differentially expressed between (1) Ph-positive and -negative patients treated with herbal paste; and (2) before and after herbal paste treatment in the Ph-positive patient group.

In the second year, Twenty-seven participants with persistent allergic rhinitis each received four acupoint herbal plaster treatments and 8 courses of acupuncture treatment over 4 weeks in the same time.

DETAILED DESCRIPTION:
This project「The oligonucleotide chip analysis for allergic rhinitis treatment in herbal plaster and acupuncture」 will be performed at Genomic Medicine Research Core Laboratory- GMRCL in Chung Gang Memorial Hospital. Allergic rhinitis patient will receive herbal plaster treatment in the first year, blood sample was attained before and after therapy. Then investigators use oligonucleotide chip to analyze the immunomodulatory effects of TCM in the treatment of allergic rhinitis. In the second year, the patient received herbal plaster and Acupuncture treatment in the same time.

Many allergic rhinitis patients accept TCM treatment here in Taiwan. According to recent journal reports, Traditional Chinese medicine performed in accordance with the principles of TCM would show significant immune-modulating effects, herbal plaster is an effective, safe and convenient treatment for allergic rhinitis. The mechanism of its efficacy needs further study. This project plan to combine the experience of clinical doctor and GMRCL Microarray for the mechanism of herbal plaster on allergic rhinitis.

Investigators study the effects of herbal plaster treatment for allergic rhinitis in the first year. And study the combine effect of herbal plaster and Acupuncture treatment in the second year. All patients during 18-45 years old were treated over a time period of 4 weeks. Patients' general well-being and several peripheral blood parameters were determined before and after the herbal plaster treatment. RNA was extracted from the blood and pooled into patient pool. Oligonucleotide chips were used to analysis the pooled RNA each year. The microarray analysis for the genomic change before and after the herbal plaster treatment or herbal plaster with Acupuncture treatment was studied .

ELIGIBILITY:
Inclusion Criteria:

* Exhibited sneezing, runny nose, and congestion for more than 9 months of the year
* Did not take medication in the previous month
* Provided written consent to enter a Chang Gung Memorial Hospital Institutional Review Board (IRB)

Exclusion Criteria:

* Sinusitis
* Nasal polyps
* unwilling or unable to complete the full course of treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Rhinitis Quality of Life Questionnaire (RQLQ) at the third week | T0: before the first acupoint herbal plaster application, T3: the third week, 24 hours after the third acupoint herbal plaster application
  RQLQ, includes 28 questions in 7 categories. The RQLQ was designed to measure the impact of rhinitis on quality of life. It considers that allergic rhinitis patients often are troubled by nasal symptoms, eye symptoms, sleep problems, emotional problems, social issues, and other symptoms.

SECONDARY OUTCOMES:
Change from baseline in Rhinitis Quality of Life Questionnaire (RQLQ) at the fourth week | T0: before the first acupoint herbal plaster application, T5: the fourth week, 24hours after the fourth acupoint herbal plaster applications
  RQLQ, includes 28 questions in 7 categories. The RQLQ was designed to measure the impact of rhinitis on quality of life. It considers that allergic rhinitis patients often are troubled by nasal symptoms, eye symptoms, sleep problems, emotional problems, social issues, and other symptoms.
Compare gene expression levels before and after a series of acupoint herbal plaster and Acupuncture treatment | 6 times in four weeks
  GeneChip Human Genome U133 Plus2 array (Affymetrix, Santa Clara, CA, USA) containing approximately 54,675 probes. Patient peripheral blood samples were obtained in 5-ml volumes at the following 6 times (T0-T5) during the study: (1) before (T0) and 24 h after the 1st (T1) acupoint herbal plaster application; (2)the third week, before (T2) and 24 h after the 3rd (T3) acupoint herbal plaster application; and (3) the fourth week, before the 4th (T4) and 24 h after the 4th (T5) acupoint herbal plaster application.
Detect serum allergen-specific IgE antibodies in patient | When patient diagnoses were confirmed by otolaryngologists (baseline). Then the ImmunoCAP Phadiatop was performed.
  ImmunoCAP Phadiatop is a blood test widely used by ENT specialists in Taiwan to detect serum allergen-specific IgE antibodies. When patient provided written consent to enter the Chang Gung Memorial Hospital Institutional Review Board (IRB)-approved human trial, Patient diagnoses were confirmed by otolaryngologists. And the ImmunoCAP Phadiatop (InVitroSight, Phadia AB, Uppsala, Sweden) was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Hen-Hong Chang, M.D., PHD, Principal Investigator — Department of Chinese Medicine, Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tai CJ, Chien LY. The treatment of allergies using Sanfujiu: A method of applying Chinese herbal medicine paste to acupoints on three peak summer days. Am J Chin Med. 2004;32(6):967-76. doi: 10.1142/S0192415X04002569. PMID 15673201
- [Background] Tai CJ, Chang CP, Huang CY, Chien LY. Efficacy of Sanfujiu to treat allergies: patient outcomes at 1 year after treatment. Evid Based Complement Alternat Med. 2007 Jun;4(2):241-6. doi: 10.1093/ecam/nel082. Epub 2006 Nov 24. PMID 17549242
- [Background] Juniper EF, Guyatt GH. Development and testing of a new measure of health status for clinical trials in rhinoconjunctivitis. Clin Exp Allergy. 1991 Jan;21(1):77-83. doi: 10.1111/j.1365-2222.1991.tb00807.x. PMID 2021881
- [Background] Benson M, Svensson PA, Carlsson B, Jernas M, Reinholdt J, Cardell LO, Carlsson L. DNA microarrays to study gene expression in allergic airways. Clin Exp Allergy. 2002 Feb;32(2):301-8. doi: 10.1046/j.1365-2222.2002.01300.x. PMID 11929497
- [Background] Shiue HS, Lee YS, Tsai CN, Hsueh YM, Sheu JR, Chang HH. Gene expression profile of patients with phadiatop-positive and -negative allergic rhinitis treated with acupuncture. J Altern Complement Med. 2010 Jan;16(1):59-68. doi: 10.1089/acm.2009.0024. PMID 20070140
- [Background] Petti FB, Liguori A, Ippoliti F. Study on cytokines IL-2, IL-6, IL-10 in patients of chronic allergic rhinitis treated with acupuncture. J Tradit Chin Med. 2002 Jun;22(2):104-11. PMID 12125480
- [Derived] Shiue HS, Lee YS, Tsai CN, Chang HH. Treatment of allergic rhinitis with acupoint herbal plaster: an oligonucleotide chip analysis. BMC Complement Altern Med. 2016 Nov 4;16(1):436. doi: 10.1186/s12906-016-1418-0. PMID 27814709